CLINICAL TRIAL: NCT00058292
Title: A Phase I Trial Combining IDEC-Y2B8 And High-Dose Beam Chemotherapy With Hematopoietic Progenitor Cell Transplant In Patients With Relapsed Or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: Radiolabeled Monoclonal Antibody Therapy and High-Dose Chemotherapy Followed By Autologous Peripheral Stem Cell Transplant in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 99H11; NU-99H11; IDEC-NU99H11
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent mantle cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Carmustine; Cytarabine; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation; ibritumomab tiuxetan

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: Carmustine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: peripheral blood stem cell transplantation; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: filgrastim — Given at a dose of 5 μg/kg, subcutaneously daily, beginning on Day 0 (stem cell transplant day) until white blood cells measure greater than 1500/ul.
  Other Names: G-CSF; granulocyte colony stimulating factor
Biological: rituximab — Intravenous infusion of 250 mg/m2 on treatment days -22 and -14 (day 0 = stem cell transplant).
Drug: Carmustine — Part of high dose BEAM chemotherapy given on study (a combination of carmustine, etoposide, cytarabine, and melphalan). Carmustine is given at a dose of 300 mg/m2 intravenous infusion over a 2 hour period on treatment day -6 (Day 0 = stem cell transplant).
  Other Names: BCNU
Drug: cytarabine — Part of high dose BEAM chemotherapy given on study (a combination of carmustine, etoposide, cytarabine, and melphalan). Cytarabine is given at a dose of 100 mg/m2 intravenous infusion over a 1 hour period, every 12 hours on treatment days -5, -4, -3, and -2, for a total of 8 doses (Day 0 = stem cell transplant).
  Other Names: Cytosar-U; Arabinosyl; Ara-C; cytosine arabinoside
Drug: etoposide — Part of high dose BEAM chemotherapy given on study (a combination of carmustine, etoposide, cytarabine, and melphalan). Etoposide is given at a dose of 100 mg/m2 intravenous infusion over a 2 hour period every 12 hours on treatment days -5, -4, -3, and -2, for a total of 8 doses (Day 0 = stem cell transplant).
  Other Names: VP-16; VP-16-213; Vepesid; Epidophylotoxin
Drug: melphalan — Part of high dose BEAM chemotherapy given on study (a combination of carmustine, etoposide, cytarabine, and melphalan). Melphalan is given at a dose of 140 mg/m2 as an intravenous infusion over a 1 hour period on treatment day -1 (Day 0 = stem cell transplant).
Procedure: peripheral blood stem cell transplantation — On day 0, a minimum of 2.0 X 106 CD34+ cells/kg unselected peripheral blood progenitor cells (PBPC) will be reinfused following institutional guidelines for the reinfusion procedure.
Radiation: yttrium Y 90 ibritumomab tiuxetan — Patients will receive 90Y2B8 at a variable dose on treatment day -14 (Day 0 = stell cell transplant). The initial dose calculated to deliver no more than 100 cGy to critical organs (liver, lung). Doses will be escalated based on cohort of enrollment.

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies such as yttrium Y90 ibritumomab tiuxetan can locate cancer cells and deliver radioactive cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining yttrium Y90 ibritumomab tiuxetan and chemotherapy with autologous stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase I trial is studying how well giving yttrium Y90 ibritumomab tiuxetan with high-dose chemotherapy followed by autologous stem cell transplant work in treating patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 ibritumomab tiuxetan, in terms of absorbed radiation to critical organs, when administered with high-dose chemotherapy followed by autologous peripheral blood stem cell transplantation in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma.
* Determine whether the residual radioactivity detected at the time of stem cell reinfusion affects the reinfused cells and delays engraftment in patients treated with this regimen.
* Determine the duration of response and survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8).

* Radioimmunotherapy: Patients receive rituximab IV followed by indium In 111 ibritumomab tiuxetan (for imaging) IV over 10 minutes on day -22. Patients then receive rituximab IV and IDEC-Y2B8 IV over 10 minutes on day -14.

Cohorts of 3-6 patients receive escalating doses of IDEC-Y2B8 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity.

* High-dose conditioning regimen: Patients receive BEAM chemotherapy comprising carmustine IV over 2 hours on day -6, etoposide IV over 2 hours twice daily and cytarabine IV over 1 hour twice daily on days -5 to -2, and melphalan IV over 1 hour on day -1.
* Autologous stem cell transplantation: Autologous peripheral blood stem cells are reinfused on day 0. Patients receive filgrastim (G-CSF) subcutaneously daily beginning on day 0 and continuing until blood counts recover.

Patients are followed at 30 days, 3 and 6 months, and then annually for 5 years.

PROJECTED ACCRUAL: A maximum of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed B-cell non-Hodgkin's lymphoma

  * Relapsed or refractory disease
  * CD20-positive disease
* Must have received at least 1 prior treatment regimen
* Complete remission with prior conventional salvage chemotherapy is allowed
* No more than 25% lymphoma in bone marrow
* No circulating malignant cells on blood smear
* No CNS involvement by lymphoma
* No HIV- or AIDS-related lymphoma

PATIENT CHARACTERISTICS:

Age

* Over 17

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3

Hepatic

* Transaminases less than 2 times normal

Renal

* Creatinine clearance greater than 50 mL/min

Cardiovascular

* LVEF at least 45%

Pulmonary

* Corrected DLCO at least 70% of predicted
* FEV_1 or FVC greater than 60%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No serious nonmalignant disease or other condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior rituximab and recovered
* No other prior murine antibodies
* No prior stem cell transplantation
* No prior radioimmunoconjugate therapy

Chemotherapy

* See Disease Characteristics
* More than 6 weeks since prior nitrosoureas or mitomycin and recovered

Endocrine therapy

* No concurrent systemic corticosteroids

Radiotherapy

* Recovered from prior radiotherapy
* No prior external beam irradiation to more than 25% of the active bone marrow

Surgery

* More than 4 weeks since prior major surgery and recovered

Other

* More than 3 weeks since prior anticancer therapy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-04; Primary Completion 2006-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of absorbed radiation to critical organs delivered with this combination of study treatments | From first study treatment until 30 days after last study treatment.
  Dose limiting toxicities observed during and up to 30 days after the last study treatment resulting in the determination of the maximum tolerated dose of absorbed radiation to critical organs delivered by Y2B8 in combination with high-dose BEAM chemotherapy with autologous mobilized peripheral blood progenitor cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jane N. Winter, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (3):
- United States (3):
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Result] Winter J, Inwards D, Spies S, et al.: Zevalin® (90YZ) doses >.5 mCi/kg may be combined with high-dose beam and autotransplant (ASCT). [Abstract] Ann Oncol 16 (Suppl 5): A-215, v100, 2005.